CLINICAL TRIAL: NCT05646264
Title: A Real World Study on the Efficacy and Safety of Agomelatin Combined With Second Generation Antipsychotics in the Treatment of Negative Symptoms in Patients With Schizophrenia
Brief Title: A Study on the Efficacy of Agomelatine Combined With Antipsychotics to Treat Negative Symptoms in Schizophrenia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Tianjin Anding Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMN202103
Record Dates: First submitted 2022-10-25; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-10

CONDITIONS: Schizophrenia; Negative Symptoms in Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — agomelatine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monotherapy group (No Intervention): Single use of second-generation antipsychotic drugs (including olanzapine, risperidone, aripiprazole, etc.)
- Joint group (Experimental): second-generation antipsychotic drugs (including olanzapine, risperidone, aripiprazole, etc.) Add Agomelatine
  Interventions: Drug: Agomelatine

INTERVENTIONS:
Drug: Agomelatine — Agomepratine is added to a second-generation antipsychotic drug (olanzapine, aripiprazole, risperidone, etc.)
  Arms: Joint group

SUMMARY:
This study is a prospective, multicenter, controlled, real world study. Patients will be randomly enrolled into the test group and the control group at a ratio of 1:1 during the screening period. The test group will choose to add Agomepratin on the basis of a second-generation antipsychotic drug (olanzapine, aripiprazole, risperidone, etc., see Annex A), and the control group will either use a second-generation antipsychotic drug (olanzapine, aripiprazole, risperidone, etc.) for 24 consecutive weeks, To explore the efficacy and safety of the second generation antipsychotic drugs combined with agomeratine regimen in the real world for negative symptoms of schizophrenic patients. Group sequential design is used as the method of interim analysis in the research process. If the research purpose is reached in advance, the research can be terminated. The study followed GRACE standards.

DETAILED DESCRIPTION:
Schizophrenia is a group of severe mental disorders of unknown etiology, with significant abnormalities in cognitive, thinking, emotional, behavioral and other aspects of mental activities, and can lead to significant occupational and social function damage. According to the relevant data of the World Health Organization, among 135 diseases or health conditions common to young people (aged 15-44), schizophrenia ranks eighth in the total disease burden, accounting for 2.6% of the total disease burden. Statistics from developed countries show that direct expenditure caused by schizophrenia accounts for 1.4% - 2.8% of total health resource expenditure. At present, there is no relevant medical economic data in China, but it is estimated that nearly 7 million people in China are suffering from schizophrenia, which causes huge medical expenditure every year, and also causes labor loss of patients and their families. Schizophrenia is still the main disease leading to mental disability at present [1].

The clinical manifestations of schizophrenia include five dimensions: positive symptoms, negative symptoms, cognitive symptoms, aggression and hostility, anxiety and depression. The existing antipsychotics (including typical and atypical antipsychotics) have a positive effect on positive symptoms, but have a poor effect on improving symptoms in other dimensions. From the perspective of prognosis, patients with non positive symptoms as the main clinical phase usually have poor prognosis. The existing evidence shows that one of the main reasons for suicide of schizophrenic patients is long-term depressive symptoms, and negative symptoms, depression and cognitive symptoms are important factors affecting the treatment outcome of patients. The treatment of negative symptoms is one of the core problems of schizophrenia at present, which still needs more exploration. At present, the treatment of negative symptoms with second-generation antipsychotics and antidepressants has been supported by some studies. However, due to the heterogeneity of antidepressants, a large number of research results are difficult to reach a unified conclusion with high evidence level. The current clinical experience believes that despite the lack of strong RCT research, the new antidepressants are well tolerated and have less side effects, which supports the use of new antidepressants in the treatment of depressive symptoms of schizophrenics.

The pathogenesis of schizophrenia is very complex. At present, the hypothesis of dopamine dysfunction plays a major role in the neurobiochemical abnormalities of schizophrenia. Carlsson et al put forward the hypothesis of dopamine neurodevelopmental defect, which believes that the core symptoms of schizophrenia are cognitive decline and negative symptoms, which is due to the lack of dopaminergic neurogenesis. In the initial state of the disease, the patients' brain has insufficient dopaminergic nerve function. When the load of the middle cerebral cortex pathway increases (puberty), it shows that the function of the dopaminergic nerve pathway is insufficient, activating the feedback regulation pathway of brain neurotransmitters, Compensatory release of dopamine leads to excessive activation of dopaminergic neural pathway in the midbrain limbic system, causing positive symptoms. With the further extension of the course of the disease and the development of the disease, this dopamine compensation mechanism is still insufficient to compensate for the dopaminergic neural function, which leads to long-term negative symptoms and cognitive dysfunction of patients.

Agomelatine is a new type of antidepressant. Its pharmacological effect is realized by activating melatonin receptor (MT1/MT2) and antagonizing 5-HT2C receptor. Agomelatine antagonizes the 5-HT2C receptor and can specifically increase the concentration of norepinephrine and dopamine in the prefrontal cortex, thereby producing antidepressant, anti anxiety and other effects. At the same time, the activation of melatonin receptor in the brain can resynchronize the circadian rhythm and biological rhythm of patients, and improve sleep rhythm disorder and sleep phase disorder caused by various reasons. At the same time, through the synergistic effect of melatonin receptor activation and 5-HT2C receptor antagonism, it can regulate the steady-state balance of neurotransmitters in the brain, especially between 5-HT and dopamine, and restore neural function. In addition, studies have shown that agomeratine has a certain role in the regeneration of hippocampal neurons and the remodeling of neural circuits [2]. An open and prospective study abroad included 27 schizophrenic patients with depressive symptoms who received a stable dose of antipsychotic drugs combined with agomeratine. The results showed that after 6 weeks of acute treatment, the depressive symptoms of the patients were significantly improved. At the same time, negative symptoms, overall psychopathology and psychosocial performance also improved significantly, while positive symptoms remained stable [3]. Subsequently, the research team further analyzed the data, which showed that after 12 weeks of treatment with agomeratine (6 weeks of acute phase+6 weeks of stable phase), the cognitive function of patients was improved (the changes in MCCB scores were statistically different). However, due to the lack of control in the experimental design, the limitation of sample number and other reasons, the research team believed that the improvement of cognitive function of patients lacked clinical significance, It is suggested to carry out research with reasonable design for further verification. In China, a single center, single blind, controlled study conducted by Jingzhou Mental Health Center in Hubei Province included 102 chronic schizophrenic patients with negative symptoms. They were randomly divided into the treatment group of argomepratin combined with risperidone (52 cases) and the treatment group of risperidone alone (50 cases). The results showed that argomepratin combined with risperidone could significantly improve the negative symptoms of patients after 6 months of treatment, Improve the quality of life of patients [4, 5].

The above clinical studies confirm that antipsychotic drugs combined with agomeratine are safe and feasible for the treatment of schizophrenia. The combined treatment has a positive effect in improving the negative symptoms and depressive symptoms of patients. Long term treatment may have the effect of improving the cognitive function of patients. However, the current clinical research sample size is small, the follow-up period is short, and the selected patients are biased, resulting in a low level of evidence. In addition, existing studies have not studied other events (such as all-cause readmission rate, suicide/self mutilation events, etc.) and the overall medical burden of patients during the treatment process, so it is difficult to form reliable evidence-based medical evidence to promote the development of clinical treatment plans for schizophrenia.

To sum up, it is proposed to carry out this prospective, multicenter, real world study of second-generation antipsychotic drugs combined with agomeratine for schizophrenia patients, aiming to further analyze the overall benefits of the combined agomeratine regimen for schizophrenia patients, and to study in detail the treatment responses of patients in the real world, and specifically analyze the effectiveness and safety of the regimen, Grasp the advantage target population and comprehensive disease burden of the program, accurately judge the application principle and medical social benefits of the program, and ultimately promote the development of clinical treatment program for schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all the following inclusion criteria to be included in this study:

  1. Male or female aged 18-65;
  2. Conform to the diagnostic criteria of schizophrenia in the International Statistical Classification of Diseases and Related Health Problems (ICD-10);
  3. 7 < PANSS positive symptom subscale score ≤ 28 (7 items score ≤ 4, that is, no more than moderate); PANSS negative symptom subscale score ≥ 24 and at least 2 of 3 core symptoms (emotional dullness, passive/indifferent social withdrawal and lack of spontaneity and fluency in conversation) ≥ 4 points;
  4. Calgary Schizophrenia Depression Scale (CDSS) score ≤ 18 (score of 9 items ≤ 2, that is, no more than moderate);
  5. According to the judgment of the researcher, the second-generation antipsychotic drugs (including olanzapine, risperidone, aripiprazole, etc.) can be used alone or added with agomeratine on the basis of them;
  6. To voluntarily participate in this study, you need to sign an informed consent form with the legal guardian at the same time.

Exclusion Criteria:

* Exclude patients who meet any of the following criteria:

  1. Combined with brain organic mental disorder;
  2. Have a history of drug abuse or drug or alcohol dependence in the past 1 year;
  3. Suffering from serious basic diseases or physical diseases or diseases that may affect the assessment (such as hearing and vision disorders);
  4. Suffering from other serious mental disorders at the same time;
  5. Serious suicide attempt;
  6. Hepatitis B virus (HBV) surface antigen positive, hepatitis C virus (HCV) antibody positive, anti human immunodeficiency virus (HIV) antibody positive or serum transaminase increased ≥ the upper limit of normal value;
  7. With mental retardation;
  8. Allergies to Agomelatine or its excipients;
  9. Pregnant women, lactating women and women of childbearing age did not take contraceptive measures;
  10. Currently participating in clinical research of other drugs or medical devices;
  11. Other antidepressants (including but not limited to SSRI and SNRI drugs) other than agomeratine should be used in combination;
  12. Accompanied by severe positive symptoms or depressive symptoms;
  13. The researcher thinks it is not suitable to be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
PANSS | 24WEEKS
  Reduction rate of total score of PANSS negative scale ≥ 20%

SECONDARY OUTCOMES:
SANS | 24WEEKS
  The change of SANS (Scale for Assessment of Negative Symptoms) total score. minimum and maximum values：0-120, lower scores mean a better outcome.
GAF | 24WEEKS
  The change of GAF (Global Assessment Function) score minimum and maximum values：0-100, higher scores mean a better outcome.
CDSS | 24WEEKS
  The change of CDSS (Calgary Depression Scale for Schizophrenia) score minimum and maximum values：0-27, lower scores mean a better outcome.

OTHER OUTCOMES:
Health Economics Indicators | 24weeks
  Utilization of health resources, total medical and economic expenses of patients during the follow-up period, including readmission, outpatient service, rehabilitation and other indicators, such as hospitalization expenses, readmission 30 days after discharge, and related outpatient/emergency care and admission times during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: yizhenghui1971@163.com Yi, M.D, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Banasr M, Soumier A, Hery M, Mocaer E, Daszuta A. Agomelatine, a new antidepressant, induces regional changes in hippocampal neurogenesis. Biol Psychiatry. 2006 Jun 1;59(11):1087-96. doi: 10.1016/j.biopsych.2005.11.025. Epub 2006 Feb 24. PMID 16499883
- [Result] Englisch S, Jung HS, Lewien A, Becker A, Nowak U, Braun H, Thiem J, Eisenacher S, Meyer-Lindenberg A, Zink M. Agomelatine for the Treatment of Major Depressive Episodes in Schizophrenia-Spectrum Disorders: An Open-Prospective Proof-of-Concept Study. J Clin Psychopharmacol. 2016 Dec;36(6):597-607. doi: 10.1097/JCP.0000000000000587. PMID 27805978